CLINICAL TRIAL: NCT04299113
Title: A Phase I Dose Escalation/Expansion Clinical Trial of Mocetinostat in Combination With Vinorelbine in Children, Adolescents and Young Adults With Refractory and/or Recurrent Rhabdomyosarcoma (RMS)
Brief Title: Mocetinostat With Vinorelbine in Children, Adolescents & Young Adults With Refractory and/or Recurrent Rhabdomyosarcoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Mirati Therapeutics Inc. (Industry); Phase One Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-000353; NCI-2019-08263 (Registry Identifier: CTRP)
Record Dates: First submitted 2020-02-10; First posted 2020-03-06 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Rhabdomyosarcoma
Keywords: Locally Advanced Rhabdomyosarcoma; Recurrent Rhabdomyosarcoma; Refractory Rhabdomyosarcoma; Unresectable Rhabdomyosarcoma
MeSH Terms: conditions — Rhabdomyosarcoma | interventions — Vinorelbine; mocetinostat; benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (vinorelbine, mocetinostat) (Experimental): Participants receive mocetinostat in combination with vinorelbine
  Interventions: Drug: Vinorelbine; Drug: Mocetinostat

INTERVENTIONS:
Drug: Vinorelbine — Given IV
  Other Names: 3'',4''-Didehydro-4''-deoxy-C''-norvincaleukoblastine, 5''-Nor-Anhydrovinblastine, 71486-22-1, Dihydroxydeoxynorvinkaleukoblastine, nor-5''-Anhydrovinblastine, vinorelbine, VINORELBINE
Drug: Mocetinostat — Given PO
  Other Names: 726169-73-9, Benzamide, N-(2-aminophenyl)-4-[[[4-(3-pyridinyl)-2-pyrimidinyl]amino]methyl]-, MG-0103, MGCD0103, MGCD0103, N-(2-aminophenyl)-4-((4-pyridin-3-ylpyrimidin-2-ylamino)methyl)benzamide

SUMMARY:
This phase I trial studies the side effects and best dose of mocetinostat when given together with vinorelbine to see how well it works in treating children, adolescents, and young adults with rhabdomyosarcoma that has spread to nearby tissues or lymph nodes and cannot be removed by surgery (locally advanced unresectable) or has spread to other places in the body (metastatic), and does not respond to treatment (refractory) or has come back (relapsed). Mocetinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as vinorelbine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving mocetinostat and vinorelbine may work better in treating children, adolescents, and young adults with rhabdomyosarcoma compared to vinorelbine alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the first cycle dose-limiting toxicities (DLTs), maximum tolerated dose (MTD), and a biologically effective and recommended phase 2 dose (RP2D) of mocetinostat administered orally three times per week for a total of 9 doses per 21 day cycle given in combination with vinorelbine on days 1, 8, 15 of 21 day cycles in subjects with refractory or recurrent rhabdomyosarcoma (RMS). (Phase 1 Dose Escalation) II. To determine the progression-free survival (PFS), defined as time from first dose of vinorelbine to tumor progression or death due to any cause, at the RP2D of mocetinostat administered orally three times per week starting on day 3 for a total of 9 doses per 21 day cycle given in combination with vinorelbine on days 1, 8, 15 of a 21 day cycle in subjects with refractory or recurrent RMS. (Expansion Cohort)

SECONDARY OBJECTIVES:

I. Safety profile of mocetinostat in combination with vinorelbine as characterized by adverse event (AE) type, severity, timing and relationship to study drugs, as well as laboratory abnormalities in the first and subsequent treatment cycles. (Phase 1 Dose Escalation) II. Pharmacokinetics (PK) of mocetinostat in plasma. (Phase 1 Dose Escalation) III. Clinical benefit rate (CBR = complete response [CR] + partial response [PR] and stable disease [SD]) of mocetinostat + vinorelbine in metastatic/refractory/unresectable RMS. (Phase 1 Dose Escalation) IV. Antitumor activity of mocetinostat + vinorelbine in refractory/recurrent RMS as measured by overall response rate (ORR), duration of response (DOR), disease control (DC), duration of disease control, as well as progression-free survival (PFS). (Phase 1 Dose Escalation) V. Pharmacodynamics of mocetinostat on molecular targets in surrogate tissue. (Phase 1 Dose Escalation and Expansion Cohort) VI. Exploratory biomarker development to enable prediction of drug toxicity, tumor response and the mechanism(s) of acquired study drug resistance. (Phase 1 Dose Escalation and Expansion Cohort) VII. Obtain RMS tissue biological samples pre-treatment and at progression to assess for differences in gene expression by next gen (generation) sequencing and ribonucleic acid (RNA) sequencing (seq). (Phase 1 Dose Escalation and Expansion Cohort) VIII. Antitumor activity of mocetinostat + vinorelbine in metastatic/refractory RMS as measured by overall response rate (ORR) and duration of response (DOR), disease control (DC), duration of disease control, as well as progression-free survival (PFS) according to Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. (Expansion Cohort) IX. Safety and tolerability of mocetinostat and vinorelbine as characterized by adverse event type, severity, timing and relationship to study drug, as well as laboratory abnormalities. (Expansion Cohort)

OUTLINE: This is a phase I, dose-escalation study of mocetinostat followed by additional studies.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved informed consent. For subjects < 18 years of age, their parents or legal guardians must sign a written informed consent. Assent, when appropriate, will be obtained according to institutional guidelines
* Have histologically or cytological confirmed diagnosis of rhabdomyosarcoma with locally advanced/unresectable, metastatic, refractory or relapsed disease who have failed standard therapy and for whom no known curative therapy exists
* Measurable disease according to RECIST version 1.1
* Prior cancer therapy: Subjects may have received any number of prior therapy regimens. In the investigator's opinion, subjects must have tolerated prior cytotoxic therapies well and have adequate bone marrow reserve. At the time of treatment initiation, at least 3 weeks must have elapsed after prior cytotoxic chemotherapy. At least 7 days must have elapsed since completion of any prior non-cytotoxic cancer therapy and any associated AEs must have resolved
* Prior radiotherapy is allowed if >= 2 weeks have elapsed for local palliative radiation therapy (XRT) (small port); >= 6 months must have elapsed if prior total body irradiation, craniospinal XRT or if > 50% radiation of the pelvis; > 6 weeks must have elapsed if other substantial bone marrow radiation (defined per principal investigator's [PI's] discretion). Subjects who have received brain irradiation must have completed whole brain radiotherapy and/or gamma knife at least 4 weeks prior to enrollment
* Subjects with controlled asymptomatic central nervous system (CNS) involvement are allowed in absence of therapy with anticonvulsants. Subjects not requiring steroids or requiring steroids at a stable dose (=< 4 mg/day dexamethasone or equivalent) for at least 2 weeks are eligible
* Resolution of all acute toxic effects (excluding alopecia) of any prior anti-cancer therapy to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (version 4.03) grade < 1 or to the baseline laboratory values as defined below
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2 in subjects >= 17 years old; or Karnofsky/Lansky > 50 in subjects < 16 years old
* Subjects age > 18 years for first cohort. Subjects must be > 12 years old for the second and subsequent cohorts
* Life expectancy of at least 3 months
* Absolute neutrophil count (ANC) >= 1000/mm^3 (>= 1.0 x 10^9/L)
* Platelets (PLT) >= 100,000/mm^3 (>= 100 x 10^9/L) (transfusion independent, defined as not receiving platelet transfusions within a 7 day period prior to screening)
* Hemoglobin > 9.0 g/dL (transfusions are allowed)
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or creatinine clearance > 60 mL/min
* Total serum bilirubin =< 1.5 x ULN; =< 5 x ULN if Gilbert's syndrome
* Liver transaminases (aspartate aminotransferase [AST]/alanine aminotransferase [ALT]) =< 2.5 x ULN; =< 5 x ULN if liver metastases are present
* Pregnancy test if female of child-bearing potential negative within 7 days of starting treatment
* Cardiac ejection fraction > 50% or shortening fraction > 28% by echocardiography (ECHO) or multigated acquisition scan (MUGA)
* Females of child-bearing potential must have a negative pregnancy test during screening and be neither breastfeeding nor intending to become pregnant during study participation. Females of childbearing potential must agree to avoid pregnancy during the study and commit to abstinence from heterosexual intercourse or agree to use two methods of birth control (one highly effective method and one additional effective method) at least 4 weeks before the start of protocol therapy, for the duration of study participation, and for 6 months after the last dose of mocetinostat
* Males with partner(s) of childbearing potential must take appropriate precautions to avoid fathering a child from the screening period until 90 days after receiving the last dose of mocetinostat. They must commit to abstinence from heterosexual intercourse or agree to use appropriate barrier contraception
* Prior to enrollment of females or males of reproductive potential, the investigator must document confirmation of the subject's understanding of the possible teratogenic effects of mocetinostat
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures

Exclusion Criteria:

* Current participation in another therapeutic clinical trial
* Symptomatic brain metastases
* History of previous cancer (non RMS), except squamous cell or basal-cell carcinoma of the skin or any in situ carcinoma that has been completely resected, which required therapy within the previous 3 years. Other low grade cancers can be reviewed and allowed at the discretion of the PI
* Incomplete recovery from any surgery (other than central venous catheter or port placement) prior to treatment
* Any of the following in the past 6 months: pericarditis, pericardial effusion, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, pulmonary embolism, deep vein thrombosis, symptomatic bradycardia, requirement for anti-arrhythmic medication
* History of prolonged corrected QT (QTc) interval (e.g., repeated demonstration of a QTc interval > 450 milliseconds, unless associated with the use of medications known to prolong the QTc interval). QTc will be calculated using the Bazett formula (RR interval = 60/heart rate; QTI corrected = QT interval/sqr[RRinterval])
* History of additional risk factors for torsade de pointes (e.g., heart failure, family history of long QT syndrome)
* Use of concomitant medications that increase or possibly increase the risk to prolong the QTc interval and/or induce torsades de pointes ventricular arrhythmia
* Females who are breastfeeding/lactating
* Known active infections (e.g., bacterial, fungal, viral including hepatitis and human immunodeficiency virus [HIV] positivity)
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study or compromise protocol objectives in the opinion of the investigator and/or the sponsor

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-05-14 (Actual); Primary Completion 2026-05-22 (Estimated); Study Completion 2027-05-22 (Estimated)

PRIMARY OUTCOMES:
To describe any dose-limiting toxicity (DLT) | 1 year
  Percentage of subjects with dose-limiting toxicities (DLTs) as assessed by NCI CTCAE (Version 4.03)
To determine the maximum tolerated dose (MTD) or highest protocol defined doses (in the absence of exceeding the MTD) | 1 year
  The MTD is the highest dose associated with first-cycle DLT in < 33% of subjects

SECONDARY OUTCOMES:
To determine the Recommended Phase 2 Dose (RP2D) for mocetinostat in combination with vinorelbine | 1 year
  The RP2D may be determined by the MTD or optimal target inhibition with an acceptable safety profile
Incidence of Adverse Events (AEs) as assessed by NCI CTCAE (Version 4.03) | 1 year
  Assess incidence of all AEs by NCI CTCAE (Version 4.03) grades 1-5
Objective Tumor Response | 2 years
  Measured using RECIST, Version 1.1
Progression Free Survival (PFS) | 2 years
  Estimated using Kaplan-Meier methodology
Disease Control (DC) | 2 years
  Proportion of subjects with a confirmed Complete Response (CR), Partial Response (PR), or Stable Disease (SD) according to RECIST v1.1
Duration of Response (DOR) | 2 years
  Measured from the first date a response is identified (either CR or PR) until the date of disease progression
Area under the Plasma Concentration versus Time Curve (AUC) of mocetinostat | 2 years
  Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums
Clearance (CL) of mocetinostat | 2 years
  Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums
Half-Life [T1/2] of mocetinostat | 2 years
  Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums
Volume of Distribution (Vd) of mocetinostat | 2 years
  Continuous variables will be summarized with means, standard deviations, medians, minimums, and maximums

CONTACTS AND LOCATIONS:
Overall Officials: Noah C. Federman, MD, Principal Investigator — University of California at Los Angeles
Locations (1):
- Rebecca Phelan, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No